CLINICAL TRIAL: NCT01926847
Title: Single Dose, Double-blind, Placebo-controlled, Single Center, Randomized Cross-over Study to Investigate Safety, Tolerability, Pharmacodynamics and Pharmacokinetic Properties of BAY63-2521 After Oral Dosing in 20 Patients With Raynaud's Phenomenon (RP)
Brief Title: Digital Flow Enhancement in Raynaud's Phenomenon With an sGC (Soluble Guanylate Cyclase) Stimulator
Acronym: DIGIT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: 16787; 2013-001899-38 (EudraCT Number)
Record Dates: First submitted 2013-08-19; First posted 2013-08-21 (Estimated); Last update posted 2014-06-16 (Estimated); Status verified 2014-06

CONDITIONS: Raynaud Disease
Keywords: Digital ischemia; Raynaud's phenomenon
MeSH Terms: conditions — Raynaud Disease | interventions — riociguat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Riociguat+Placebo (Experimental): Randomization order 1: first single oral dose of 2 mg BAY63-2521, then matching placebo
  Interventions: Drug: Riociguat (Adempas, BAY63-2521); Drug: Placebo
- Placebo+Riociguat (Experimental): Randomization order 2: first matching placebo, then single oral dose of 2 mg BAY63-2521
  Interventions: Drug: Riociguat (Adempas, BAY63-2521); Drug: Placebo

INTERVENTIONS:
Drug: Riociguat (Adempas, BAY63-2521)
Drug: Placebo

SUMMARY:
Patients with Raynaud's phenomenon suffer from painful attacks triggered by stress or cold causing acute lowering of blood flow through the digits. In this trial the safety and efficacy as well as the effect of one dose of the sGC stimulator Riociguat on digital blood flow will be measured during a cold exposure test in patients suffering from Raynaud's phenomenon. Measurements of two periods will be compared: in one period the patient will be given active drug and in the other period a placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from Raynaud's phenomenon diagnosed at least ≥1 year before beginning of the study of the following origin:

  * idiopathic (primary)
  * limited cutaneous Scleroderma associated
  * diffuse cutaneous Scleroderma associated
  * mixed connective tissue disease associated

Exclusion Criteria:

* Patients taking medication interfering with the digital flow measurement such as calcium channel blockers (CCB), phosphodiesterase 5 (PDE5) inhibitors, endothelin receptor antagonists (ERA), Nitrates
* Smokers
* Systolic blood pressure (SBP) below 105mmHg at rest

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-10; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | 5 weeks
Blood pressure | 5 weeks
Pulse rate | 5 weeks
Incidence of participants showing changes during clinical laboratory and hematology assessment | From baseline to 5 weeks
Plasma concentration at 2 h after riociguat administration | After 2 hours
Placebo corrected change in digital blood flow at room temperature, measured by Laser Doppler Perfusion Imaging | At baseline and after 2h
Placebo corrected change in digital blood flow during cold exposure, measured by Laser Doppler Perfusion Imaging | At baseline and after 2h

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Cologne, North Rhine-Westphalia, Germany